CLINICAL TRIAL: NCT01648452
Title: A Phase I/II Study of the NT-501 Intraocular Implant Releasing Ciliary Neurotrophic Factor (CNTF) in Participants With CNGB3 Achromatopsia
Brief Title: CNTF Implants for CNGB3 Achromatopsia
Acronym: CNTF-CNGB3-1
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Paul A. Sieving, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120167; 12-EI-0167
Record Dates: First submitted 2012-07-20; First posted 2012-07-24 (Estimated); Results first posted 2014-02-25 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-09

CONDITIONS: Eye Disease; Achromatopsia
Keywords: Achromatopsia; Ciliary Neurotrophic Factor; CNTF
MeSH Terms: conditions — Eye Diseases; Color Vision Defects

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- NT-501 CNTF-releasing implant (Experimental): Ocular implantation of a NT-501 CNTF-releasing capsule (20 ng/day) in one eye (the study eye) at baseline
  Interventions: Biological: NT-501 CNTF-releasing implant

INTERVENTIONS:
Biological: NT-501 CNTF-releasing implant — 20 ng/day released into the eye

SUMMARY:
Background:

* Achromatopsia is an inherited condition that causes vision loss because cells in the retina do not work properly. It causes loss of acuity, sensitivity to light, and loss of color vision. There are no effective treatments for achromatopsia.
* Four genes currently are known to cause achromatopsia. One of these, the cyclic nucleotide-gated channel beta 3 (CNGB3) gene, is the cause in about 50 percent of people.
* CNTF is a natural chemical found in the body that promotes survival and function of nerve cells. CNTF has been shown to be effective in treating retinal disease in animals and can slow vision loss.
* CNTF has also been studied in over 250 people with retinal disease other than achromatopsia. In these studies, a CNTF implant was placed into the eye during a simple surgery. The implant releases CNTF inside the eye, near the retina. These studies suggested that a CNTF implant might help vision in some eye diseases.

Objectives:

* To learn whether a CNTF implant is safe for people with CNGB3 achromatopsia.
* To learn whether CNTF can improve visual acuity or color vision, and whether it may reduce sensitivity to light in people with CNGB3 achromatopsia.

Eligibility:

You may be able to take part in this study if you:

* Are at least 18 years old.
* Test positive for mutations in the CNGB3 gene and have no mutations in another achromatopsia gene.
* Have 20/100 vision or worse in at least one eye.
* Are not pregnant or nursing.

Design:

* To determine if you can take part, we will ask about your medical history and do a physical examination and an eye examination. Blood and urine samples will be taken.
* This study requires 11 visits to the National Eye Institute over 3 years.
* One visit will be for the implant surgery. The implant will be placed in one eye only.
* Study visits will take place 1 day after implant surgery, and again 1 week later and 1 month, 3 months, 6 months, 1 year, 1.5 years and 3 years later. These visits will help us evaluate the safety and benefit of the implant on your eye.
* At the 3 year visit, you can choose to keep the CNTF implant in your eye, or you can have us remove it.

DETAILED DESCRIPTION:
Objective: The objective of this study is to evaluate the safety of ocular NT-501 device with encapsulated NT-201 cells releasing Ciliary Neurotrophic Factor (CNTF) to the retina of participants affected with CNGB3 achromatopsia.

Study Population: Five participants affected with CNGB3 achromatopsia will be enrolled, with one eye treated per participant.

Design: This is a Phase I/II, prospective, single-center study. One eye of each participant will receive a vitreous NT-501 device implant releasing CNTF. The study will be completed once the final participant has received three years of follow-up.

Outcome Measures: The primary outcome is the number and severity of adverse events and systemic and ocular toxicities at six months post-implantation. Additional safety of ocular CNTF implants in participants with CNGB3 achromatopsia will be determined from assessment of retinal function, ocular structure and occurrence of adverse events at all time points. Secondary outcomes include changes in visual function including visual acuity and color vision, electroretinogram (ERG) responses, and retinal imaging with optical coherence tomography (OCT).

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the following inclusion criteria must be met, where applicable.

* Participant must be 18 years of age or older.
* Participant must carry two alleles for CNGB3 gene mutations and no cyclic nucleotide-gated channel alpha 3 (CNGA3) sequence variations as confirmed in a Clinical Laboratory Improvement Amendments (CLIA)-certified laboratory.
* Participant must understand and sign the protocol informed consent.
* Both female participants of childbearing potential and male participants able to father children must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse, or must agree to use contraception during the first six months following implantation. Acceptable forms of contraception include:hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring), intrauterine device, barrier methods (diaphragm, condom) with spermicide, or surgical sterilization (tubal ligation).

Exclusion Criteria:

A participant is not eligible if any of the following exclusion criteria are present.

* Participant has a history of other ocular disease likely to contribute significantly to visual loss (e.g., optic neuropathy, glaucoma, uveitis, or other retinal disease).
* Participant is judged by the investigator as not sufficiently healthy to safely undergo ophthalmic surgery.
* Participant is on anticoagulant therapy that cannot be safely stopped peri-operatively at the implant procedure. Patients on warfarin will always be excluded. Patients on aspirin will be asked to stop the medication at least seven days prior to the surgery (when not contraindicated by the underlying medical condition). The stoppage period for other anticoagulant medications is based on the best clinical judgment of the investigator surgeon and is variable depending on the patient's medical condition and the type of medication.
* Participant has had diagnosis or treatment of a malignancy (excluding non-melanoma skin cancer) within the previous five years.
* Participant has received investigational treatment in another clinical study related to an ocular condition in the last six months.
* Participant is pregnant, lactating or planning to become pregnant in the first six months following implantation.

Study Eye Eligibility Criteria:

The participant must have at least one eye meeting all inclusion criteria and none of the exclusion criteria listed below.

Study Eye Inclusion Criteria:

The study eye must have a best-corrected Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity letterscore of ≤ 53 (i.e., ≤ 20/100). The visual acuity from the first baseline visit (Baseline 1) will be used for eligibility determination in case of a change in visual acuity at the second baseline visit (Baseline 2).

Study Eye Exclusion Criteria:

* The study eye has a choroidal nevus or ocular neoplasm with potential risk for malignant transformation.
* The study eye is judged by the investigator, based on history or examination findings, as high-risk for retinal detachment, vitreous hemorrhage, infection, or uveitis.
* The study eye has lens, cornea, or other media opacities precluding adequate visualization and testing of the retina.
* The study eye has undergone intraocular surgery within 12 months prior to enrollment.

Study Eye Selection Criteria in Cases of Bilateral Disease:

* As this is a genetic condition that usually affects both eyes to a similar degree, if both eyes of a participant meet the study eye eligibility criteria and have comparable visual acuity, the study eye will be selected at the investigator's medical judgment after consultation with the participant.
* In case of an eye with lower visual acuity, that eye will be selected as the study eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-07; Primary Completion 2013-03 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Sieving, MD, PhD, Principal Investigator — National Eye Institute (NEI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kohl S, Baumann B, Broghammer M, Jagle H, Sieving P, Kellner U, Spegal R, Anastasi M, Zrenner E, Sharpe LT, Wissinger B. Mutations in the CNGB3 gene encoding the beta-subunit of the cone photoreceptor cGMP-gated channel are responsible for achromatopsia (ACHM3) linked to chromosome 8q21. Hum Mol Genet. 2000 Sep 1;9(14):2107-16. doi: 10.1093/hmg/9.14.2107. PMID 10958649
- [Background] Wissinger B, Gamer D, Jagle H, Giorda R, Marx T, Mayer S, Tippmann S, Broghammer M, Jurklies B, Rosenberg T, Jacobson SG, Sener EC, Tatlipinar S, Hoyng CB, Castellan C, Bitoun P, Andreasson S, Rudolph G, Kellner U, Lorenz B, Wolff G, Verellen-Dumoulin C, Schwartz M, Cremers FP, Apfelstedt-Sylla E, Zrenner E, Salati R, Sharpe LT, Kohl S. CNGA3 mutations in hereditary cone photoreceptor disorders. Am J Hum Genet. 2001 Oct;69(4):722-37. doi: 10.1086/323613. Epub 2001 Aug 30. PMID 11536077
- [Background] Kohl S, Baumann B, Rosenberg T, Kellner U, Lorenz B, Vadala M, Jacobson SG, Wissinger B. Mutations in the cone photoreceptor G-protein alpha-subunit gene GNAT2 in patients with achromatopsia. Am J Hum Genet. 2002 Aug;71(2):422-5. doi: 10.1086/341835. Epub 2002 Jun 20. PMID 12077706
- [Result] Zein WM, Jeffrey BG, Wiley HE, Turriff AE, Tumminia SJ, Tao W, Bush RA, Marangoni D, Wen R, Wei LL, Sieving PA. CNGB3-achromatopsia clinical trial with CNTF: diminished rod pathway responses with no evidence of improvement in cone function. Invest Ophthalmol Vis Sci. 2014 Sep 9;55(10):6301-8. doi: 10.1167/iovs.14-14860. PMID 25205868
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2012-EI-0167.html

RESULTS

PARTICIPANT FLOW:
Groups:
- NT-501 CNTF-releasing Implant: Participants received an ocular implantation of a NT-501 CNTF-releasing capsule (20 ng/day) in one eye (the study eye) at baseline.
Period: Overall Study
Arm/Group | NT-501 CNTF-releasing Implant
Started | 5
Completed | 5 (One participant was explanted due to an adverse event. Remainder kept implant at study completion.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.6 (11.37)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events at Six Months Post-Implantation
Description: The primary outcome is the total number of adverse events reported within six months post-implantation.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 10

2. Primary Outcome: Number of Severe Adverse Events at Six Months Post-Implantation
Description: The number of severe adverse events reported within six months post-implantation.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 1

3. Primary Outcome: Number of Ocular Adverse Events at Six Months Post-Implantation
Description: The number of eye-related adverse events reported within six months post-implantation.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 9

4. Primary Outcome: Number of Non-Ocular Adverse Events at Six Months Post-Implantation
Description: The number of non eye-related adverse events reported within six months post-implantation.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 1

5. Secondary Outcome: Number of Adverse Events at All Time Points Post-Implantation
Description: The total number of adverse events reported from Day 1 post-implantation through study completion at Year 3.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 15

6. Secondary Outcome: Number of Severe Adverse Events at All Time Points Post-Implantation
Description: The total number of severe adverse events reported from Day 1 post-implantation through study completion at Year 3.
  Although there were two serious adverse events (SAEs) reported during the study, only one event's severity was classified as "severe."
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 1

7. Secondary Outcome: Number of Ocular Adverse Events at All Time Points Post-Implantation
Description: The total number of eye-related adverse events reported from Day 1 post-implantation through study completion at Year 3.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 11

8. Secondary Outcome: Number of Non-Ocular Adverse Events at All Time Points Post-Implantation
Description: The total number of non eye-related adverse events reported from Day 1 post-implantation through study completion at Year 3.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: Adverse Events
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
Adverse Events | 4

9. Secondary Outcome: Number of Participants Who Experienced an Improvement in Visual Acuity of Greater Than 0.3 logMAR (Logarithm of the Minimum Angle of Resolution) Post-Implantation in the Study Eye.
Description: Improvement of visual acuity was assessed on both the study and control eyes. Visual acuity was measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) protocol. Acuity is measured as letters read on an ETDRS eye chart and the letters read equate to Snellen measurements. For example, if a participant reads between 84 and 88 letters, the equivalent Snellen measurement is 20/20. .
  The LogMAR scale [expressed as the (decadic) logarithm of the minimum angle of resolution (range from +1.00 to -0.30)] converts the geometric sequence of a traditional chart to a linear scale. It measures VA loss; positive values indicate vision loss, whereas negative values denote normal or better VA. A lower LogMAR value indicates better VA. For example, a visual acuity of 20/20 corresponds to a logMAR value of zero (0), and a visual acuity of 20/100 corresponds to a LogMAR value of 0.7.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
participants | 0

10. Secondary Outcome: Number of Participants Who Experienced an Improvement in Visual Acuity of Greater Than 0.3 logMAR (Logarithm of the Minimum Angle of Resolution) Post-Implantation in the Untreated Control Eye.
Description: as for outcome 9
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | Untreated Control Eye
Number analyzed (Participants) | 5
participants | 0

11. Secondary Outcome: Number of Participants Who Experienced an Increase in Either the Rod or Cone Electroretinogram (ERG) Responses of More Than 75% Post-Implantation in the Study Eye.
Description: Full-ﬁeld ERGs were recorded according to International Society of Clinical Electrophysiology of Vision Standards (ISCEV).
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
participants | 0

12. Secondary Outcome: Number of Participants Who Experienced an Increase in Either the Rod or Cone Electroretinogram (ERG) Responses of More Than 75% Post-Implantation in the Untreated Control Eye.
Description: as for outcome 11
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | Untreated Control Eye
Number analyzed (Participants) | 5
participants | 0

13. Secondary Outcome: Number of Participants Who Experienced an Improvement in Color Discrimination and/or Matching Post-Implantation in the Study Eye.
Description: Color hue discrimination was tested by the Nagel anomaloscope, American Optical Hardy Rand Rittler (AOHRR) color plates, and a low vision version of the Cambridge Color Test (LvCCT) implemented on a ViSaGe System (Cambridge Research Systems Ltd., Rochester, UK) using custom-written software. Hardy Rand Rittler testing followed the guidelines accompanying the test and administered under a Macbeth Lamp at 300 lux.
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | NT-501 CNTF-releasing Implant
Number analyzed (Participants) | 5
participants | 0

14. Secondary Outcome: Number of Participants Who Experienced an Improvement in Color Discrimination and/or Matching Post-Implantation in the Untreated Control Eye.
Description: as for outcome 13
Time Frame: Day 1, Week 1, Week 4, Week 12, Week 24, Week 52, Week 78, Week 156 post-implantation
Measure: Number; unit: participants
Arm/Group | Untreated Control Eye
Number analyzed (Participants) | 5
participants | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected at all time points until study completion (up to Week 156 post-implantation).
Description: The primary outcome is the number and severity of adverse events and systemic and ocular toxicities within six months post-implantation.
Groups:
- NT-501 CNTF-releasing Implant Events ≤ 6 Months Post-implant: Participants received an ocular implantation of a NT-501 CNTF-releasing capsule (20 ng/day) in one eye (the study eye) at baseline. The events listed reflect the primary outcome endpoint of adverse events reported within 6 months post-implantation.
- NT-501 CNTF-releasing Implant Events > 6 Months Post-implant: Participants received an ocular implantation of a NT-501 CNTF-releasing capsule (20 ng/day) in one eye (the study eye) at baseline. The events listed are adverse events reported after the primary outcome endpoint of 6 months post-implantation.
Arm/Group | NT-501 CNTF-releasing Implant Events ≤ 6 Months Post-implant | NT-501 CNTF-releasing Implant Events > 6 Months Post-implant
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/5
Other Adverse Events (participants affected / at risk) | 5/5 | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-501 CNTF-releasing Implant Events ≤ 6 Months Post-implant (N=5) | NT-501 CNTF-releasing Implant Events > 6 Months Post-implant (N=5)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Retinal Detachment (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NT-501 CNTF-releasing Implant Events ≤ 6 Months Post-implant (N=5) | NT-501 CNTF-releasing Implant Events > 6 Months Post-implant (N=5)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Delayed Dark Adaptation (Eye disorders) | 4 (4) | 0 (0) — The event coded to a MedDRA v16 Preferred Term of Night Blindness but the verbatim Lower Level Terminology is delayed dark adaptation. As the MedDRA term may misrepresent participants as being blind, the verbatim event will be utilized, not MedDRA.
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Vitreous detachment (Eye disorders) | 1 (1) | 0 (0)
Vitritis (Eye disorders) | 2 (2) | 0 (0)
Shoulder Operation (Surgical and medical procedures) | 0 (0) | 1 (1)
Lenticular Opacities (Eye disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Uterine operation (Surgical and medical procedures) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes